CLINICAL TRIAL: NCT02271347
Title: An Open-Label, Multicenter Study of the Safety and Anti Viral Activity of Brincidofovir (BCV, CMX001) for Ebola Virus Disease
Acronym: CMX
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended Development Program
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX001-205
Record Dates: First submitted 2014-10-07; First posted 2014-10-22 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2014-10

CONDITIONS: Ebola Virus
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMX001 (Experimental): CMX001 administered as initial dose of 200mg then 100mg BIW for a total of 5 doses.
  Interventions: Drug: CMX001

INTERVENTIONS:
Drug: CMX001 — CMX001 administered as initial dose of 200mg then 100mg BIW for a total of 5 doses.
  Other Names: Brincidofovir

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Brincidofovir (BCV) when administered as an initial 200mg dose followed by 100mg twice weekly (BIW) for a total of 5 doses.

ELIGIBILITY:
Inclusion Criteria:

* Positive for Ebola virus RNA in plasma
* Subject must be able to ingest, absorb, and tolerate oral medication
* Subject must be willing to use adequate contraception during their participation

Exclusion Criteria:

-

Ages: 2 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability. | 4 weeks